CLINICAL TRIAL: NCT01359150
Title: A Randomized, Double Blind, Placebo Controlled Phase 2 Study To Assess The Immune Response Following Administration Of Influenza And Pneumococcal Vaccines To Subjects With Rheumatoid Arthritis Receiving Cp-690,550 Or Placebo Cp-690,550 With And Without Background Methotrexate
Brief Title: A Study To Assess the Immune Response Following Administration Of Influenza and Pneumococcal Vaccines To Subjects With Rheumatoid Arthritis Receiving CP-690,550 Or Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3921129
Record Dates: First submitted 2011-05-11; First posted 2011-05-24 (Estimated); Results first posted 2013-03-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group 1: 10 mg BID CP-690,550 (100 subjects). (Experimental): CP-690,550 will be administered for 4 weeks, vaccines will be administered at week 4. CP-690,550 will then continue for another 5 weeks at which point the immune response will be evaluated.
  Interventions: Drug: CP-690,550
- Treatment Group 2:Placebo CP-690,550 (100 subjects). (Placebo Comparator): Placebo will be administered for 4 weeks, vaccines will be administered at week 4. Placebo will then continue for another 5 weeks at which point the immune response will be evaluated.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CP-690,550 — Treatment Group 1: 10 mg BID CP-690,550 (100 subjects). Strata 1: 10 mg BID CP-690,550 on background methotrexate (50 subjects); Strata 2: 10 mg BID CP-690,550 monotherapy (50 subjects).
  Arms: Treatment Group 1: 10 mg BID CP-690,550 (100 subjects).
Drug: placebo — Placebo CP-690,550 (100 subjects). Strata 1: Placebo CP-690,550 on background methotrexate (50 subjects); Strata 2: Placebo CP-690,550 monotherapy (50 subjects). Influenza and pneumococcal vaccines will be administered to all subjects
  Arms: Treatment Group 2:Placebo CP-690,550 (100 subjects).

SUMMARY:
A Randomized, Double Blind, Placebo Controlled Phase 2 Study To assess the Immune Response Following Administration of Influenza and Pneumococcal Vaccines to Subjects with Rheumatoid Arthritis receiving CP-690,550 with and Without background Methotrexate

ELIGIBILITY:
Inclusion Criteria:

* The subject must meet the American College of Rheumatology (ACR) classification criteria for the diagnosis of RA by satisfying at least four of the seven criteria.
* The subject must have active disease at both screening and baseline

Exclusion Criteria:

* History of any documented influenza or pneumococcal infection within the last 3 months.
* Receipt of any vaccine within 1 month prior to the initial study drug administration (CP-690,550 or placebo CP-690,550).
* If a subject has received an influenza vaccine within 6 months or a pneumococcal vaccine within 5 years of initial study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- United States (48):
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, Paradise Valley, Arizona
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Fair Oaks, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Roseville, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Trumbull, Connecticut
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Port Richey, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Zephyrhills, Florida
  - Pfizer Investigational Site, Morton Grove, Illinois
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Vernon Hills, Illinois
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Cumberland, Maryland
  - Pfizer Investigational Site, Leominster, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Bingham Farms, Michigan
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Binghamton, New York
  - Pfizer Investigational Site, Olean, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Rocky Mount, North Carolina
  - Pfizer Investigational Site, Minot, North Dakota
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Mesquite, Texas
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Vancouver, Washington
  - Pfizer Investigational Site, Clarksburg, West Virginia
- Poland (6):
  - Pfizer Investigational Site, Cieszyn
  - Pfizer Investigational Site, Kościan
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Torun
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Winthrop KL, Silverfield J, Racewicz A, Neal J, Lee EB, Hrycaj P, Gomez-Reino J, Soma K, Mebus C, Wilkinson B, Hodge J, Fan H, Wang T, Bingham CO 3rd. The effect of tofacitinib on pneumococcal and influenza vaccine responses in rheumatoid arthritis. Ann Rheum Dis. 2016 Apr;75(4):687-95. doi: 10.1136/annrheumdis-2014-207191. Epub 2015 Mar 20. PMID 25795907
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921129&StudyName=A%20Study%20To%20Assess%20the%20Immune%20Response%20Following%20Administration%20Of%20Influenza%20and%20Pneumococcal%20Vaccines%20To%20Subjects%20with%20Rheumatoid%20Arthriti

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 + Influenza and Pneumococcal Vaccine: CP-690,550 10 milligram (mg) tablet orally twice daily up to Day 64, with or without background Methotrexate therapy as per local standard prescribing practice. Participants were vaccinated on Day 29 with influenza and pneumococcal vaccine based on standard practice.
- Placebo + Influenza and Pneumococcal Vaccine: Placebo matched to CP-690,550 10 mg tablet orally twice daily up to Day 64, with or without background Methotrexate therapy as per local standard prescribing practice. Participants were vaccinated on Day 29 with influenza and pneumococcal vaccine based on standard practice.
Period: Overall Study
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine
Started | 112 | 111
Completed | 105 | 106
Not Completed | 7 | 5
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 4 | 3
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine | Total
Number analyzed (Participants) | 112 | 111 | 223
Age Continuous [Mean (Standard Deviation); unit: years] | 52.7 (10.4) | 52.2 (11.1) | 52.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 90 | 171
  Male | 31 | 21 | 52
Number of Participants With Background (BG) Methotrexate (MTX) use [Number; unit: participants]
  With Background MTX use | 62 | 62 | 124
  Without Background MTX use | 50 | 49 | 99

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Satisfactory Humoral Response to the Pneumococcal Vaccine at Visit 3 (Day 64)
Description: Satisfactory humoral response to the pneumococcal vaccine was defined as greater than or equal to (>=) 2 fold increase in antibody concentrations from vaccination baseline (Day 29) in at least 6 of 12 pneumococcal antigens (1, 3, 4, 5, 6B, 7F, 9V, 14, 19A, 19F, 23F, 18C). Data was stratified by the background methotrexate use.
Time Frame: Day 64 (End of Study [EOS])
Population: Evaluable immunogenicity population:eligible,randomized participants;who met rheumatoid arthritis disease activity criteria;received vaccination as scheduled and >=80% study drug;had pre and post-vaccination blood draw;complete set of assay results;had no major protocol violations.n=participants evaluable at specified categories for each arm group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine
Number analyzed (Participants) | 102 | 98
percentage of participants
  Regardless MTX use (n=102,98) | 45.1 [35.224 to 55.264] | 68.4 [58.196 to 77.394]
  With BG MTX use (n=57,55) | 31.6 [19.905 to 45.243] | 61.8 [47.726 to 74.591]
  Without BG MTX use (n=45,43) | 62.2 [46.541 to 76.232] | 76.7 [61.369 to 88.245]

2. Primary Outcome: Percentage of Participants With Satisfactory Humoral Response to the Seasonal Influenza Vaccine at Visit 3 (Day 64)
Description: Satisfactory humoral response to the influenza vaccine was defined as >= 4 fold increase in antibody titers from vaccination baseline (Day 29) in at least 2 of 3 influenza antigens (B, H1N1, H3N2). Data was stratified by the background methotrexate use.
Time Frame: Day 64 (EOS)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine
Number analyzed (Participants) | 102 | 98
percentage of participants
  Regardless MTX use (n=102,98) | 56.9 [46.682 to 66.634] | 62.2 [51.885 to 71.844]
  With BG MTX use (n=57,55) | 50.9 [37.29 to 64.37] | 58.2 [44.106 to 71.345]
  Without BG MTX use (n=45,43) | 64.4 [48.78 to 78.132] | 67.4 [51.456 to 80.924]

3. Secondary Outcome: Percentage of Participants Who Responded to Each of the 12 Pneumococcal Antigens
Description: Response to the pneumococcal vaccine (seroconversion) was defined as >= 2 fold increase in antibody concentrations from vaccination baseline (Day 29) in each of the 12 pneumococcal antigens (1, 3, 4, 5, 6B, 7F, 9V, 14, 19A, 19F, 23F, 18C). Data was stratified by the background methotrexate use.
Time Frame: Day 64 (EOS)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine
Number analyzed (Participants) | 102 | 98
percentage of participants
  Regardless MTX use, 1 (n=102,98) | 59.8 [49.63 to 69.393] | 69.4 [59.265 to 78.302]
  Regardless MTX use, 14 (n=102,98) | 52 [41.844 to 61.961] | 61.2 [50.849 to 70.903]
  Regardless MTX use, 18C (n=102,98) | 59.8 [49.63 to 69.393] | 70.4 [60.338 to 79.205]
  Regardless MTX use, 19A (n=102,98) | 32.4 [23.424 to 42.337] | 46.9 [36.778 to 57.289]
  Regardless MTX use, 19F (n=102,98) | 35.3 [26.086 to 45.38] | 56.1 [45.732 to 66.133]
  Regardless MTX use, 23F (n=102,98) | 40.2 [30.607 to 50.37] | 58.2 [47.766 to 68.054]
  Regardless MTX use, 3 (n=102,98) | 38.2 [28.787 to 48.386] | 54.1 [43.714 to 64.196]
  Regardless MTX use, 4 (n=102,98) | 58.8 [48.644 to 68.477] | 65.3 [55.02 to 74.64]
  Regardless MTX use, 5 (n=102,98) | 28.4 [19.938 to 38.218] | 38.8 [29.097 to 49.151]
  Regardless MTX use, 6B (n=102,98) | 36.3 [26.982 to 46.386] | 54.1 [43.714 to 64.196]
  Regardless MTX use, 7F (n=102,98) | 58.8 [48.644 to 68.477] | 65.3 [55.02 to 74.64]
  Regardless MTX use, 9V (n=102,98) | 45.1 [35.224 to 55.264] | 58.2 [47.766 to 68.054]
  With BG MTX use, 1 (n=57,55) | 57.9 [44.084 to 70.857] | 61.8 [47.726 to 74.591]
  With BG MTX use, 14 (n=57,55) | 47.4 [33.985 to 61.035] | 56.4 [42.322 to 69.696]
  With BG MTX use, 18C (n=57,55) | 49.1 [35.63 to 62.71] | 58.2 [44.106 to 71.345]
  With BG MTX use, 19A (n=57,55) | 19.3 [10.047 to 31.911] | 40 [27.023 to 54.093]
  With BG MTX use, 19F (n=57,55) | 28.1 [16.973 to 41.543] | 49.1 [35.354 to 62.929]
  With BG MTX use, 23F (n=57,55) | 24.6 [14.127 to 37.761] | 49.1 [35.354 to 62.929]
  With BG MTX use, 3 (n=57,55) | 24.6 [14.127 to 37.761] | 49.1 [35.354 to 62.929]
  With BG MTX use, 4 (n=57,55) | 52.6 [38.965 to 66.015] | 56.4 [42.322 to 69.696]
  With BG MTX use, 5 (n=57,55) | 28.1 [16.973 to 41.543] | 29.1 [17.63 to 42.898]
  With BG MTX use, 6B (n=57,55) | 29.8 [18.429 to 43.403] | 47.3 [33.653 to 61.196]
  With BG MTX use, 7F (n=57,55) | 49.1 [35.63 to 62.71] | 56.4 [42.322 to 69.696]
  With BG MTX use, 9V (n=57,55) | 33.3 [21.401 to 47.065] | 49.1 [35.354 to 62.929]
  Without BG MTX use, 1 (n=45,43) | 62.2 [46.541 to 76.232] | 79.1 [63.958 to 89.956]
  Without BG MTX use, 14 (n=45,43) | 57.8 [42.15 to 72.343] | 67.4 [51.456 to 80.924]
  Without BG MTX use, 18C (n=45,43) | 73.3 [58.055 to 85.396] | 86 [72.068 to 94.702]
  Without BG MTX use, 19A (n=45,43) | 48.9 [33.703 to 64.226] | 55.8 [39.875 to 70.922]
  Without BG MTX use, 19F (n=45,43) | 44.4 [29.644 to 60.003] | 65.1 [49.073 to 78.992]
  Without BG MTX use, 23F (n=45,43) | 60 [44.331 to 74.302] | 69.8 [53.875 to 82.818]
  Without BG MTX use, 3 (n=45,43) | 55.6 [39.997 to 70.356] | 60.5 [44.41 to 75.023]
  Without BG MTX use, 4 (n=45,43) | 66.7 [51.05 to 79.999] | 76.7 [61.369 to 88.245]
  Without BG MTX use, 5 (n=45,43) | 28.9 [16.366 to 44.315] | 51.2 [35.465 to 66.695]
  Without BG MTX use, 6B (n=45,43) | 44.4 [29.644 to 60.003] | 62.8 [46.725 to 77.025]
  Without BG MTX use, 7F (n=45,43) | 71.1 [55.685 to 83.634] | 76.7 [61.369 to 88.245]
  Without BG MTX use, 9V (n=45,43) | 60 [44.331 to 74.302] | 69.8 [53.875 to 82.818]

4. Secondary Outcome: Percentage of Participants Who Responded to Each of the 3 Influenza Antigens
Description: Response to the influenza vaccine (seroconversion) was defined as >= 4 fold increase in antibody titers from vaccination baseline (Day 29) in each of 3 influenza antigens (B, H1N1, H3N2). Data was stratified by the background methotrexate use.
Time Frame: Day 64 (EOS)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine
Number analyzed (Participants) | 102 | 98
percentage of participants
  Regardless MTX use, B (n=102,98) | 38.2 [28.787 to 48.386] | 52 [41.712 to 62.243]
  Regardless MTX use, H1N1 (n=102,98) | 60.8 [50.62 to 70.305] | 63.3 [52.925 to 72.781]
  Regardless MTX use, H3N2 (n=102,98) | 60.8 [50.62 to 70.305] | 69.4 [59.265 to 78.302]
  With BG MTX use, B (n=57,55) | 35.1 [22.915 to 48.869] | 41.8 [28.655 to 55.894]
  With BG MTX use, H1N1 (n=57,55) | 52.6 [38.965 to 66.015] | 58.2 [44.106 to 71.345]
  With BG MTX use, H3N2 (n=57,55) | 57.9 [44.084 to 70.857] | 65.5 [51.419 to 77.763]
  Without BG MTX use, B (n=45,43) | 42.2 [27.657 to 57.85] | 65.1 [49.073 to 78.992]
  Without BG MTX use, H1N1 (n=45,43) | 71.1 [55.685 to 83.634] | 69.8 [53.875 to 82.818]
  Without BG MTX use, H3N2 (n=45,43) | 64.4 [48.78 to 78.132] | 74.4 [58.828 to 86.481]

5. Secondary Outcome: Percentage of Participants With Protective Antibody Titers to the Seasonal Influenza Vaccine
Description: Seroprotection was defined as achieving protective antibody titers to the influenza vaccine as measured by a hemagglutination inhibition (HAI) assay titer of >= 1:40 in at least 2 of 3 influenza antigens (B, H1N1, H3N2). Data was stratified by the background methotrexate use.
Time Frame: Day 64 (EOS)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine
Number analyzed (Participants) | 102 | 98
percentage of participants
  Regardless MTX use (n=102,98) | 76.5 [67.043 to 84.305] | 91.8 [84.547 to 96.41]
  With BG MTX use (n=57,55) | 64.9 [51.131 to 77.085] | 92.7 [82.413 to 97.983]
  Without BG MTX use (n=45,43) | 91.1 [78.779 to 97.525] | 90.7 [77.865 to 97.407]

6. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Anti-Pneumococcal Antibody Levels to Each of the 12 Pneumococcal Antigens Above Vaccination Baseline Values (Day 29)
Description: Geometric mean fold rises (GMFRs) for the 12 pneumococcal antigens (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) from pre-vaccination (Day 29) to Day 64 (Day 35 post-vaccination) were computed using the logarithmically transformed assay results. Confidence intervals (CIs) for GMFR are back transformations of a CI based on the Student t-distribution for the mean logarithm of the titers. Data was stratified by the background methotrexate use.
Time Frame: Day 64 (EOS)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine
Number analyzed (Participants) | 102 | 98
fold rise
  Regardless MTX use, 1 (n=89,92) | 4.75 [3.61 to 6.24] | 6.83 [4.94 to 9.46]
  Regardless MTX use, 14 (n=101,96) | 2.68 [2.19 to 3.28] | 3.90 [3.05 to 4.99]
  Regardless MTX use, 18C (n=101,98) | 3.10 [2.52 to 3.81] | 4.82 [3.76 to 6.18]
  Regardless MTX use, 19A (n=102,98) | 1.80 [1.56 to 2.08] | 2.34 [1.99 to 2.75]
  Regardless MTX use, 19F (n=102,95) | 2.04 [1.71 to 2.42] | 2.89 [2.40 to 3.49]
  Regardless MTX use, 23F (n=102,98) | 2.00 [1.64 to 2.44] | 2.81 [2.34 to 3.36]
  Regardless MTX use, 3 (n=101,94) | 2.11 [1.76 to 2.54] | 2.79 [2.31 to 3.38]
  Regardless MTX use, 4 (n=96,89) | 3.10 [2.49 to 3.86] | 5.13 [3.94 to 6.67]
  Regardless MTX use, 5 (n=101,98) | 1.72 [1.50 to 1.97] | 2.27 [1.91 to 2.70]
  Regardless MTX use, 6B (n=102,98) | 1.90 [1.61 to 2.24] | 2.56 [2.12 to 3.10]
  Regardless MTX use, 7F (n=102,97) | 3.19 [2.59 to 3.93] | 4.06 [3.27 to 5.04]
  Regardless MTX use, 9V (n=102,98) | 2.27 [1.85 to 2.55] | 3.16 [2.59 to 3.86]
  With BG MTX use, 1 (n=49,53) | 3.92 [2.77 to 5.54] | 4.51 [3.00 to 6.77]
  With BG MTX use, 14 (n=56,54) | 2.37 [1.84 to 3.04] | 2.85 [2.19 to 3.72]
  With BG MTX use, 18C (n=57,55) | 2.64 [2.05 to 3.41] | 3.23 [2.45 to 4.26]
  With BG MTX use, 19A (n=57,55) | 1.51 [1.30 to 1.74] | 2.08 [1.67 to 2.59]
  With BG MTX use, 19F (n=57,53) | 1.92 [1.51 to 2.44] | 2.29 [1.88 to 2.79]
  With BG MTX use, 23F (n=57,55) | 1.66 [1.32 to 2.07] | 2.34 [1.88 to 2.91]
  With BG MTX use, 3 (n=56,54) | 1.78 [1.39 to 2.27] | 2.43 [1.90 to 3.12]
  With BG MTX use, 4 (n=53,50) | 2.92 [2.22 to 3.85] | 3.27 [2.51 to 4.25]
  With BG MTX use, 5 (n=57,55) | 1.62 [1.35 to 1.95] | 1.99 [1.59 to 2.50]
  With BG MTX use, 6B (n=57,55) | 1.60 [1.37 to 1.88] | 2.24 [1.79 to 2.81]
  With BG MTX use, 7F (n=57,55) | 2.38 [1.89 to 2.98] | 3.46 [2.57 to 4.64]
  With BG MTX use, 9V (n=57,55) | 1.87 [1.53 to 2.29] | 2.72 [2.08 to 3.54]
  Without BG MTX use, 1 (n=40,39) | 6.01 [3.85 to 9.37] | 12.04 [7.34 to 19.74]
  Without BG MTX use, 14 (n=45,42) | 3.14 [2.25 to 4.37] | 5.85 [3.81 to 8.99]
  Without BG MTX use, 18C (n=44,43) | 3.80 [2.70 to 5.35] | 8.05 [5.37 to 12.08]
  Without BG MTX use, 19A (n=45,43) | 2.27 [1.75 to 2.94] | 2.72 [2.13 to 3.47]
  Without BG MTX use, 19F (n=45,42) | 2.19 [1.68 to 2.85] | 3.88 [2.78 to 5.43]
  Without BG MTX use, 23F (n=45,43) | 2.54 [1.81 to 3.58] | 3.55 [2.63 to 4.78]
  Without BG MTX use, 3 (n=45,40) | 2.61 [1.98 to 3.44] | 3.37 [2.49 to 4.55]
  Without BG MTX use, 4 (n=43,39) | 3.32 [2.31 to 4.79] | 9.15 [5.85 to 14.29]
  Without BG MTX use, 5 (n=44,43) | 1.86 [1.50 to 2.29] | 2.68 [2.04 to 3.52]
  Without BG MTX use, 6B (n=45,43) | 2.36 [1.73 to 3.21] | 3.04 [2.19 to 4.21]
  Without BG MTX use, 7F (n=45,42) | 4.62 [3.23 to 6.60] | 5.02 [3.65 to 6.90]
  Without BG MTX use, 9V (n=45,43) | 2.63 [2.03 to 3.41] | 3.83 [2.82 to 5.19]

7. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Anti-Influenza Antibody Levels to Each of the Influenza Antigens Above Vaccination Baseline Values (Day 29)
Description: GMFRs for the 3 influenza antigens (B, H1N1, H3N2) from pre-vaccination (Day 29) to Day 64 (Day 35 post-vaccination) were computed using the logarithmically transformed assay results. CIs for GMFR are back transformations of a CI based on the Student t-distribution for the mean logarithm of the titers. Data was stratified by the background methotrexate use.
Time Frame: Day 64 (EOS)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine
Number analyzed (Participants) | 102 | 98
fold rise
  Regardless MTX use, B (n=102,98) | 2.95 [2.32 to 3.75] | 3.90 [3.06 to 4.97]
  Regardless MTX use, H1N1 (n=102,98) | 6.04 [4.59 to 7.95] | 9.50 [6.76 to 13.35]
  Regardless MTX use, H3N2 (n=102,98) | 7.11 [5.18 to 9.75] | 9.06 [6.61 to 12.44]
  With BG MTX use, B (n=57,55) | 2.84 [2.02 to 3.98] | 3.11 [2.27 to 4.26]
  With BG MTX use, H1N1 (n=57,55) | 4.90 [3.43 to 7.00] | 7.54 [4.80 to 11.85]
  With BG MTX use, H3N2 (n=57,55) | 5.69 [3.88 to 8.34] | 6.04 [4.18 to 8.73]
  Without BG MTX use, B (n=45,43) | 3.11 [2.20 to 4.40] | 5.20 [3.57 to 7.57]
  Without BG MTX use, H1N1 (n=45,43) | 7.88 [5.13 to 12.10] | 12.76 [7.56 to 21.53]
  Without BG MTX use, H3N2 (n=45,43) | 9.43 [5.52 to 16.09] | 15.25 [9.06 to 25.66]

8. Secondary Outcome: Geometric Mean Concentrations (GMC) of Anti-Pneumococcal Antibody
Description: Antibody geometric mean concentration (GMC) for 12 pneumococcal antigens (1, 3, 4, 5, 6B, 7F, 9V, 14, 19A, 19F, 23F, 18C) as measured by geometric mean of three independent determinations of the antibody response of that antigen. GMC and corresponding 2-sided 95% confidence intervals (CI) were evaluated.
Time Frame: Day 64 (EOS)
Population: Evaluable immunogenicity population:eligible,randomized participants;who met rheumatoid arthritis disease activity criteria;received vaccination as scheduled and >=80% study drug;had pre and post-vaccination blood draw;complete set of assay results;had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram/milliliter (mcg/mL)
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine
Number analyzed (Participants) | 102 | 98
microgram/milliliter (mcg/mL)
  1 | 1.81 [1.32 to 2.48] | 3.27 [2.34 to 4.58]
  14 | 5.24 [3.85 to 7.12] | 6.40 [4.63 to 8.84]
  18C | 2.53 [1.95 to 3.29] | 4.60 [3.48 to 6.09]
  19A | 5.21 [4.15 to 6.54] | 8.57 [6.86 to 10.70]
  19F | 2.59 [1.93 to 3.47] | 3.09 [2.28 to 4.19]
  23F | 2.41 [1.86 to 3.11] | 3.55 [2.78 to 4.55]
  3 | 0.66 [0.52 to 0.86] | 1.11 [0.86 to 1.43]
  4 | 0.72 [0.54 to 0.97] | 1.07 [0.77 to 1.48]
  5 | 4.05 [3.23 to 5.09] | 5.79 [4.60 to 7.30]
  6B | 2.99 [2.34 to 3.83] | 4.75 [3.71 to 6.07]
  7F | 3.28 [2.42 to 4.45] | 4.37 [3.36 to 5.67]
  9V | 2.61 [2.11 to 3.23] | 4.06 [3.29 to 5.01]

9. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-Influenza Antibody
Description: Antibody geometric mean titer (GMT) for 3 influenza antigens antigens (B, H1N1, H3N2) as measured by geometric mean of three independent determinations of the antibody response of that antigen. GMT and corresponding 2-sided 95% confidence intervals (CI) were evaluated.
Time Frame: Day 64 (EOS)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine
Number analyzed (Participants) | 102 | 98
titer
  B | 33.39 [25.61 to 43.54] | 50.74 [39.82 to 64.64]
  H1N1 | 86.40 [64.35 to 116.0] | 221.5 [161.4 to 304.0]
  H3N2 | 132.3 [97.65 to 179.1] | 244.0 [184.6 to 322.5]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 + Influenza and Pneumococcal Vaccine | Placebo + Influenza and Pneumococcal Vaccine
Serious Adverse Events (participants affected / at risk) | 4/112 | 1/111
Other Adverse Events (participants affected / at risk) | 17/112 | 17/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 + Influenza and Pneumococcal Vaccine (N=112) | Placebo + Influenza and Pneumococcal Vaccine (N=111)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 + Influenza and Pneumococcal Vaccine (N=112) | Placebo + Influenza and Pneumococcal Vaccine (N=111)
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 8
Urinary tract infection (Infections and infestations) | 3 | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 5 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.